CLINICAL TRIAL: NCT01337037
Title: Modified Video-assisted Thoracoscopic Surgery (VATS) Lobectomy for Early-stage Non-small Cell Lung Cancer (NSCLC)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Collaborators: Shanghai Zhongshan Hospital (Other); West China Hospital (Other); Sun Yat-sen University (Other); The First Hospital of Jilin University (Other); Central South University (Other); Jiangsu Cancer Institute & Hospital (Other); Beijing Friendship Hospital (Other); Xuanwu Hospital, Beijing (Other); Peking University (Other); Fujian Provincial Hospital (Other); Fuzhou General Hospital (Other); Beijing Haidian Hospital (Other); Fuzhou Pulmonary Hospital of Fujian (Other)
Responsible Party: Principal Investigator, Jun Wang, prof. Dr., Peking University People's Hospital
Other Study IDs: PHTD2010
Record Dates: First submitted 2011-04-06; First posted 2011-04-18 (Estimated); Last update posted 2015-01-27 (Estimated); Status verified 2015-01

CONDITIONS: Lung Cancer
Keywords: video-assisted thoracic surgery; Lung cancer; lobectomy
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- standard VATS group: patients undergo standard VATS lobectomy using non-modified equipments,without limits of staples
  Interventions: Procedure: Standard VATS lobectomy
- modified equipments group: patients undergo VATS lobectomy with modified VATS lobectomy equipments designed designed according to the experience of chinese lobectomy surgery: Lobectomy Equipments Pack (Manufacturer B.J.ZH.F.Panther Medical Equipment Co.,Ltd.).
  Interventions: Device: VATS lobectomy using modified equipments
- less staples group: patients undergo VATS lobectomy with at most 4 staples used.
  Interventions: Procedure: VATS lobectomy using less staples
- open group: patients undergo lobectomy by thoracotomy approach
  Interventions: Procedure: Open lobectomy

INTERVENTIONS:
Device: VATS lobectomy using modified equipments — the procedure of this group is the same with standard VATS lobectomy group.the VATS surgical equipments used in the group are designed according to the experience of chinese lobectomy surgery. All the patent applications of the surgical equipments are granted. proprietor of the patents is Jun Wang, head of Department of Thoracic surgery of people's hospital, peking university.
  Details of the modified equipments: Lobectomy Equipments Pack (Manufacturer B.J.ZH.F.Panther Medical Equipment Co.,Ltd.) consists of 8 basic surgical equipments, which are crafoord dissecting and ligature forcep, Yankauer suction tube, mixter dissecting and ligature forceps(long),mixter dissecting and ligature forceps(short), atraumatic-grip aorta-aneurysma clamp with toothing De Bakey, De Bakey atraumatic-grip vascular forcep, Bozemann tite grip needle holder, Winter placenta and ovum forcep.
  Groups: modified equipments group
Procedure: VATS lobectomy using less staples — VATS lobectomy with at most 4 staples used, aimed at reduced hospital cost.This procedure is similar with the standard VATS lobectomy procedure without staples limits. The lobar vessels and bronchus are stapled. However, the interlobar fissures should be deal with electronic cautery, harmonic scalpel,or suturing.
  Groups: less staples group
Procedure: Standard VATS lobectomy — VATS lobectomy without new equipments and limitation of staples, same with the current procedure of VATS lobectomy performed in thoracic departments of Peking university people's hospital and the Collaborators. All procedures were conducted under general anesthesia with double lumen intubation. The thoracoscope was introduced through 7th or 8th intercostals space on the mid-axillaries line. The 4 cm long utility incision was made on the 4th or 5th intercostals space anterior axillary's line without rib-spreading. A third retraction incision located on the 7th or 8th intercostals space sub-scapular line. The surgeon stands on the ventral side of patient using an electrocautery hook and a suction device through the utility incision. Anatomic lobectomy was performed with systemic mediastinal lymph node dissection for lung cancer patients.
  Groups: standard VATS group
Procedure: Open lobectomy — standard lobectomy procedure by thoracotomy approach
  Groups: open group

SUMMARY:
The purpose of this study is to modify the surgical technique of VATS (video-assisted thoracoscopic surgery) lobectomy for early-stage non-small cell lung cancer.

DETAILED DESCRIPTION:
VATS (video-assisted thoracoscopic surgery) lobectomy is a relatively new minimally invasive surgical treatment for early-stage non-small cell lung cancer (NSCLC), associated with low morbidity and mortality and effective oncologic results over the standard thoracotomy. However, this surgical procedure has not spread widely in china for several reasons. First , VATS surgery cost more than thoracotomy for thoracoscopic staples; second, the procedure of VATS lobectomy may be more difficult in china as the lack of VATS surgical equipments adjusted for smaller thoracic cavity of chinese, and more common adhesive and calcified lymph nodes due to infection and tuberculosis; Third, the surgical levels of VATS lobectomy are far from equal in china, and the Continuing Medical Education training programs of thoracoscopic surgery seem to be less efficient without major criterion.

The purpose of this study is to modify the surgical technique of VATS (video-assisted thoracoscopic surgery) lobectomy for early-stage non-small cell lung cancer, to examine the feasibility of VATS lobectomy performed by less staples, and to evaluate the feasibility of VATS lobectomy performed by modified surgical equipments designed according to the experience of chinese lobectomy surgery, and to generate a chinese standard operative procedure of VATS lobectomy for technique learning and spread. The investigators will intend to recruit 250 patients each group, for 4 groups. Group A(open group) will undergo radical lobectomy via thoracotomy approach. Group B(standard VATS group) will undergo lobectomy via standard VATS approach introduced. Group C(less staples group) will undergo lobectomy via VATS approach with staples limitation. Group D(modified equipments group) will undergo lobectomy via VATS approach using VATS surgical equipments designed according to the experience of chinese lobectomy surgery. The investigators will compare two groups of patients as followed: A vs. B, B vs. C, B vs. D.

ELIGIBILITY:
Inclusion Criteria:

1. clinically diagnosed with stage I to stage II peripheral non-small cell lung cancer suitable for lobectomy.
2. signed informed consent from patient or legal representative, and allowed adequate follow-up.
3. operators must have experience of VATS lobectomy for more than 50 cases.

Exclusion Criteria:

1. pregnant or breastfeeding women.
2. severe complications or infections.
3. no prior chemotherapy or radiotherapy for this malignancy.
4. medical history of mediastinal or hilar lymphadenopathy.
5. current participation in another study involving an investigational device or drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: in hospital patients
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2011-04; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Operative time | 6 weeks after surgery.
  For modified equipments group, if the operative time is significantly less than stand VATS group, the equipments is considered as feasible.
Survival time | 5 years
  overall survival rate(1-year, 3-year,5-year)will be analysed by the survival times of the follow-up patients.
Hospital cost | 6 weeks after surgery.
  less staples group vs.standard VATS group

SECONDARY OUTCOMES:
Quality of life | 1 year
  measured by Zubrod-ECOG-WHO score
Pain Scale Evaluation | 6 weeks after surgery
  measured by Visual analog scale (VAS)
Blood loss | 3 months after surgery
  to evaluate the blood loss volume as followed:open group vs. standard VATS group; modified equipments group vs. standard VATS group; less staples group vs.standard VATS group.
Postoperative mortality | 3 months after surgery
  to evaluate the postoperative mortality as followed: open group vs. standard VATS group; modified equipments group vs. standard VATS group; less staples group vs.standard VATS group.
Conversion rate | 6 weeks after surgery
  For modified equipments group, if conversion rates is not significantly different with stand VATS group, and success rate is over 90%, VATS lobectomy is considered as feasible.
Disease-free survival time | 5 years after surgery
  overall Disease-free survival rate(1-year, 3-year,5-year)will be analysed by the survival times of the follow-up patients.
Postoperative morbidity | 3 months after surgery
  to evaluate the postoperative morbidity above as followed: open group vs. standard VATS group; modified equipments group vs. standard VATS group; less staples group vs.standard VATS group.
Postoperative drainage duration | 3 months after surgery
  to evaluate the postoperative drainage duration as followed: open group vs. standard VATS group; modified equipments group vs. standard VATS group; less staples group vs.standard VATS group.
Postoperative hospital stay | 3 months after surgery
  to evaluate the postoperative hospital stay above as followed: open group vs. standard VATS group; modified equipments group vs. standard VATS group; less staples group vs.standard VATS group.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Wang, MD, Study Director — Department of Thoracic Surgery, Center for Mini-invasive Thoracic Surgery, People's Hospital, Peking University
Locations (14):
- China (14):
  - Department of Thoracic Surgery, Center for Mini-invasive Thoracic Surgery, People's Hospital, Peking University, Beijing, Beijing Municipality
  - Beijing Haidian hospital, Beijing, Beijing Municipality
  - Department of Thoracic Surgery，Beijing Friendship Hospital, Beijing, Beijing Municipality
  - Department of Thoracic Surgery，Peking University School of Oncology, Beijing, Beijing Municipality
  - Department of Thoracic Surgery，Xuanwu Hospital Capital Medical University, Beijing, Beijing Municipality
  - Department of Thoracic Surgery，Fuzhou Pulmonary Hospital of Fujian, Fuzhou, Fujian
  - Department of Thoracic Surgery, Fuzhou General Hospital of Nanjing Military Command, Fuzhou, Fujian
  - Department of Thoracic Surgery，Fujian Provincial Hospital, Fuzhou, Fujian
  - Department of Oncologic Surgery, Sun Yat-sen Univisity Cancer Center, Guangzhou, Guangdong
  - Department of Thoracic Surgery, the second Xiangya Hospital of Central South University, Changsha, Hunan
  - Department of Thoracic Surgery, Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - Department of Thoracic Surgery，Jilin University Norman Bethune Hospital, Changchun, Jilin
  - Department of Thoracic Surgery，Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality
  - Department of Thoracic Surgery, West China Hospital,Sichuan University, Chengdu, Sichuan

REFERENCES:
- [Background] Li Yun, Wang Jun, Sui Xi-zhao, et al. Operative technique optimization in completely thoracoscopic lobectomy: Peking University experience: CHINESE JOURNAL OF THORACIC AND CARDIOVASCULAR SURGERY 2010;26(5).